CLINICAL TRIAL: NCT06992947
Title: Does the British Columbia Farmers' Market Nutrition Coupon Program Improve the Diet Quality and Food Security of Parents and Children With Lower Incomes? A Dose-response, Pragmatic Randomized Controlled Trial
Brief Title: Impact of Healthy Food Subsidies on Diet Quality and Food Security
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); British Columbia Farmers' Market Nutrition Coupon Program (Other); BC Association of Farmers' Markets (Unknown)
Responsible Party: Principal Investigator, Dana Lee Olstad, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB24-1774; 195904 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Food Insecurity
Keywords: Randomized controlled trial; diet quality; food insecurity; low-income; healthy food subsidy; adults; children; parental shielding; dose-response; farmers market

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded to group assignment but will be blinded to the study objectives. Community partners who distribute coupons and vendors who redeem coupons at farmers' markets will be blinded to group assignment. Researchers who collect and analyze the data will not be involved in delivering the intervention and thus will remain blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SUBSIDY-2 (Experimental): Participants in this group will receive 16 weeks of coupons valued at $54/household/week, which is two times higher than the usual FMNCP subsidy. The subsidy will be provided in the form of coupons that can be used to purchase healthy foods at BC farmers' markets, including vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs. Participants will also be invited to participate in nutrition skill-building activities (e.g. cooking and gardening classes) offered by community partners. Participation in these activities is optional, which is consistent with the existing FMNCP.
  Interventions: Other: Healthy food subsidy: $54/household/week; Other: Nutrition skill-building
- SUBSIDY-3 (Experimental): Participants in this group will receive 16 weeks of coupons valued at $81/household/week, which is three times higher than the usual FMNCP subsidy. The subsidy will be provided in the form of coupons that can be used to purchase healthy foods at BC farmers' markets, including vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs. Participants will also be invited to participate in nutrition skill-building activities (e.g. cooking and gardening classes) offered by community partners. Participation in these activities is optional, which is consistent with the existing FMNCP.
  Interventions: Other: Healthy food subsidy: $81/household/week; Other: Nutrition skill-building
- SUBSIDY-Usual (Active Comparator): Participants in this group will receive 16 weeks of coupons valued at $27/household/week, which is the usual FMNCP subsidy. The subsidy will be provided in the form of coupons that can be used to purchase healthy foods at BC farmers' markets, including vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs. Participants will also be invited to participate in nutrition skill-building activities (e.g. cooking and gardening classes) offered by community partners. Participation in these activities is optional, which is consistent with the existing FMNCP.
  Interventions: Other: Healthy food subsidy: $27/household/week; Other: Nutrition skill-building

INTERVENTIONS:
Other: Healthy food subsidy: $27/household/week — Participants receive 16 weeks of coupons valued at $27/week to purchase healthy foods at BC farmers' markets. Eligible foods include vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs.
  Arms: SUBSIDY-Usual
Other: Healthy food subsidy: $54/household/week — Participants receive 16 weeks of coupons valued at $54/week to purchase healthy foods at BC farmers' markets. Eligible foods include vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs.
  Arms: SUBSIDY-2
Other: Healthy food subsidy: $81/household/week — Participants receive 16 weeks of coupons valued at $81/week to purchase healthy foods at BC farmers' markets. Eligible foods include vegetables, fruits, dairy, meat, poultry, fish, eggs, nuts, vegetable and fruit plants, honey and herbs.
  Arms: SUBSIDY-3
Other: Nutrition skill-building — Participants are eligible, but not required, to attend optional nutrition skill-building activities (e.g. cooking and gardening classes).

SUMMARY:
The British Columbia Farmers' Market Nutrition Coupon Program (FMNCP) provides lower-income households with coupons to purchase healthy foods at farmers' markets. This pragmatic randomized controlled trial (RCT) will examine the effectiveness and cost-effectiveness of two higher subsidies for healthy food ($54/weeek or $81/week), compared to the usual FMNCP healthy food subsidy ($27/week), on the diet quality (primary outcome), food insecurity, and other health-related outcomes of 276 parent-child dyads with lower incomes. 276 parent-child dyads who are enrolled in the FMNCP will be randomly assigned to one of the three subsidy arms. Participants will receive 16 weeks of coupons that can be redeemed for up to 20 weeks. Outcomes will be assessed in one parent (18-64 years) and child (6-17 years) from each household pre-, mid- and post-intervention.

DETAILED DESCRIPTION:
Background: The British Columbia Farmers' Market Nutrition Coupon Program (FMNCP) is a healthy eating initiative designed to facilitate access to nutritious food for lower-income households. The program provides households with 16 weeks of coupons valued at $27/week to purchase healthy foods at BC farmers' markets, including fruits, vegetables, dairy, meat, poultry, fish, eggs, nuts, fruit and vegetable plants, honey and herbs. The expectation is that individuals will purchase and consume healthier foods when they are financially supported to do so, and that their overall well-being and health will improve as a result.

In a prior randomized controlled trial (RCT) in adults, the investigators found that the FMNCP did not improve adults' diet quality; however, it did reduce household food insecurity by 79%. It is hypothesized that parents in the prior RCT predominantly used their subsidies to feed their children and that higher subsidies are needed to ensure both parents and children benefit. A novel dose-response RCT among parent-child dyads is essential to examine how variations in subsidy amounts affect distinct outcomes among parents and children.

This pragmatic RCT will examine the effectiveness and cost-effectiveness of two higher subsidies for healthy food, compared to the usual FMNCP healthy food subsidy, on the diet quality (primary outcome), food insecurity, and other health-related outcomes of 276 parent-child dyads with lower incomes. The primary outcome is overall diet quality post-intervention. Secondary outcomes mid- and post-intervention include: 1) Other dietary outcomes: overall diet quality (mid-intervention only), diet quality components, food purchasing, intake of ultra-processed foods; 2) Food insecurity: food insecurity status and severity, nutrition security, parental shielding; and 3) Self-reported health-related outcomes: mental well-being, sense of community, perceived stress, perceived health, food literacy, BMI.

Methods: In this single-blind, three-arm, parallel-group pragmatic RCT, 276 parent-child dyads in lower-income households will be randomized to receive the usual FMNCP healthy food subsidy ($27/week) or a subsidy that is two ($54/week) or three times ($81/week) higher. Participants will receive 16 weeks of coupons that can be redeemed for up to 20 weeks. Outcomes will be assessed in one parent (18-64 years) and one child (6-17 years) from each household pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons). Dietary intake will be collected via two 24-hour dietary recalls using the Automated Self-Administered 24-hour Dietary Recall at each time point to assess diet quality. Foods purchased with coupons will be assessed by analyzing pictures taken by participants. Food insecurity and other health-related outcomes will be assessed using validated self-reported instruments. Mixed effects regression will assess the effects of the interventions, relative to the usual food subsidy, on outcomes in parents and children. A full incremental analysis will quantify the cost-effectiveness ratios of the three healthy food subsidies.

ELIGIBILITY:
Inclusion Criteria:

* Meet existing FMNCP-specific annual household income eligibility cut-offs that account for the local cost of living
* Have 2-5 members in the household, specifically with a parent 18-64 years and a child 6-17 years. If there are multiple eligible individuals, the parent who is the primary food shopper and the youngest child will be enrolled.
* Parent-child dyads must reside together ≥5 days/week
* Are the only dyad in their household participating in the study
* Have access to the internet and a camera
* Able to communicate in English or have someone to translate

Exclusion Criteria:

* Trying to conceive, pregnant or breastfeeding
* Participating in other trials that might interfere with the intervention
* Reside in a facility that provides meals (e.g., shelter, long-term care) or where they cannot prepare meals (e.g., hotel)
* Anticipate being outside of their community for >2 consecutive weeks during the study
* Expect to move to a non-FMNCP community during the study
* Expect a significant change in their household income or composition during the study

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 538 (Actual)
Dates: Start 2025-06-07 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Overall Diet Quality in Parents | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in diet quality by Healthy Eating Food Index-2019 scores in parents. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-80. A higher score indicates a higher diet quality.
Overall Diet Quality in Children | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in diet quality by Healthy Eating Food Index-2019 scores in children. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-80. A higher score indicates a higher diet quality.

SECONDARY OUTCOMES:
Overall Diet Quality in Parents | Assessed pre- and mid-intervention (i.e., after 8 weeks of coupons have been distributed)
  Difference between intervention groups and SUBSIDY-Usual in diet quality by Healthy Eating Food Index-2019 scores in parents. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-80. A higher score indicates a higher diet quality.
Overall Diet Quality in Children | Assessed pre- and mid-intervention (i.e., after 8 weeks of coupons have been distributed)
  Difference between intervention groups and SUBSIDY-Usual in diet quality by Healthy Eating Food Index-2019 scores in children. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-80. A higher score indicates a higher diet quality.
Diet Quality Component Scores in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in diet quality component scores by Healthy Eating Food Index-2019 in parents. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-5 or 0-10 depending on the component. A higher score indicates higher intake of the specified component, with the exception of moderation components (higher score indicates lower intake).
Diet Quality Component Scores in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in diet quality component scores by Healthy Eating Food Index-2019 in children. Dietary intake will be collected via two 24-hour dietary recalls at each time point to calculate diet quality. Scores can range from 0-5 or 0-10 depending on the component. A higher score indicates higher intake of the specified component, with the exception of moderation components (higher score indicates lower intake).
Percent Energy from Ultra-Processed Foods in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in percent of energy consumed from ultra-processed foods in parents. Two dietary recalls will be used to calculate percent energy from ultra-processed foods using the NOVA classification.
Percent Energy from Ultra-Processed Foods in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in percent of energy consumed from ultra-processed foods in children. Two dietary recalls will be used to calculate percent energy from ultra-processed foods using the NOVA classification.
Household Food Insecurity Status | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in household food insecurity status (food secure or food insecure) in the past 30 days. Health Canada's 18-item Household Food Security Survey Module will be used to assess whether households experienced food insecurity in the past 30 days. If there are no affirmative responses to any of the 18 items households will be classified as food secure; otherwise they will be classified as food insecure (i.e., if there are 1 or more affirmative responses).
Parental Shielding | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in parental shielding (shielded or not shielded) in the past 30 days. Health Canada's 18-item Household Food Security Survey will be used to assess parental shielding in the past 30 days. Shielding exists when there are one or more affirmative responses on the 10-item adult scale, but there are no affirmative responses on the 8-item child scale.
Household Food Insecurity Severity | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in experiences of household food insecurity in the past 30 days. Health Canada's 18-item Household Food Security Survey Module will be used to assess experiences of marginal (1 affirmative response on the adult and/or child scale), moderate (2-5 affirmative responses on the adult scale or 2-4 affirmative responses on the child scale), and severe (≥6 affirmative responses on the adult scale or ≥5 affirmative responses on the child scale) household food insecurity in the past 30 days.
Household Nutrition Security | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in nutrition security scores. Gretchen Swanson Centre's Nutrition Security Survey will be used to assess experiences of nutrition security at a household level. The scale will be modified to the past 30 days. The 4-item survey uses a 5-point Likert scale. Each item is scored from 0=always to 4=never. Total scores are reported as a mean of the item scores. A higher score indicates a greater degree of household nutrition security.
Proportion of Coupons Spent on Foods Classified as Minimally Processed, Culinary, Ingredients, Processed, and Ultra-processed | Assessed each time participants purchase food using FMNCP coupons from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Difference between intervention groups and SUBSIDY-Usual in proportion of coupons (based on dollar value) spent on foods classified as minimally processed, culinary, ingredients, processed, and ultra-processed. Participants will take photos of the foods purchased with coupons and report the number of coupons used to purchase the items. Foods purchased will be classified using the NOVA food classification system: minimally processed, culinary, ingredients, processed, and ultra-processed.
Proportion of Coupons Spent on Foods Classified as Very Poor, Poor, Fair, Good and Excellent Choice | Assessed each time participants purchase food using FMNCP coupons from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Difference between intervention groups and SUBSIDY-Usual in proportion of coupons (based on dollar value) spent on foods classified as very poor, poor, fair, good, and excellent choice. Participants will take photos of the foods purchased with coupons and report the number of coupons used to purchase the items. Foods purchased will be classified using the Canadian Food Scoring System as very poor, poor, fair, good, and excellent choice.
Proportion of Coupons Spent on Foods Classified as Sell Most, Sell Sometimes and Do Not Sell | Assessed each time participants purchase food using FMNCP coupons from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Difference between intervention groups and SUBSIDY-Usual in proportion of coupons (based on dollar value) classified as sell most, sell sometimes, and do not sell. Participants will take photos of the foods purchased with coupons and report the number of coupons used to purchase the items. Foods purchased will be classified using the British Columbia Ministry of Health Standards: sell most, sell sometimes, and do not sell.
Mental Well-Being in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in Warwick-Edinburgh Mental Well-Being Scale scores (range 14-70) in the past 2 weeks in parents. A higher score indicates better mental well-being.
Mental Well-Being in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in Stirling Children's Wellbeing Scale scores (range 12-60) in the past 2 weeks in children. A higher score indicates better mental well-being.
Sense of Community in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in Brief Sense of Community Scale scores in parents. Responses range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 8-40. A higher score indicates a stronger sense of community.
Perceived Stress in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in perceived stress in parents. The 14-item Perceived Stress Scale-10 will be used to assess perceived stress over the past month in parents. Scores can range from 0-40. Higher scores indicate higher perceived stress.
Perceived Stress in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in perceived stress in children. The 14-item Perceived Stress Scale for Children will be used to assess perceived stress in children over the previous week. Scores can range from 0-39. Higher scores indicate higher perceived stress.
Food Literacy in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in food literacy scores in parents. Food literacy is measured via the 23-item Canadian Food Literacy Measure. Scores can range from 20-115. Higher scores indicate higher food literacy.
Self-Rated Health in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in perceived health in parents. Single-item question from the Canadian Community Health Survey used to self-rate current health as poor, fair, good, very good or excellent.
Self-Rated Health in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in perceived health in children. Single-item question from the Canadian Community Health Survey used to self-rate current health as poor, fair, good, very good or excellent.
Body Mass Index in Parents | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in BMI in parents. Self-reported height (cm or inches) and weight (kg or lbs) used to calculate BMI (kg per meter squared).
Body Mass Index Z-Scores in Children | Assessed pre-, mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Difference between intervention groups and SUBSIDY-Usual in BMI in children. Self-reported height (cm or inches) and weight (kg or lbs) used to calculate BMI (kg per meter squared) z-scores .

OTHER OUTCOMES:
Coupon Receipt | Assessed bi-weekly from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Receipt of FMNCP coupons is verified using records from community partners indicating dates when coupons were distributed to participants.
Coupon Redemption | Assessed each time participants purchase food using FMNCP coupons from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Farmers' market vendors return all coupons that were redeemed to the researchers. Coupons have serial numbers that are linked to study participants. Participants also take photos of foods purchased with coupons and report the number of coupons used to purchase the items.
Nutrition Skill-Building Activity Attendance | Assessed based on written records recorded from pre- to post-intervention (i.e., when the farmers' market a household shops at closes for the season)
  Attendance to nutrition skill-building activities is verified using records from community partners indicating dates when participants attended nutrition skill-building activities.
Subgroup Analyses by Sex | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on BMI differed by sex
Subgroup Analyses by Gender | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by gender
Subgroup Analyses by Ethnicity | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by ethnicity
Subgroup Analyses by Household Size | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by household size
Subgroup Analyses by Household Food Insecurity Status at Baseline | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by household food insecurity status at baseline
Subgroup Analyses According to the Average Value of FMNCP Coupons Redeemed Prior to Dietary Recalls | Assessed mid- (i.e., after 8 weeks of coupons have been distributed) and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed according to the average value of FMNCP coupons redeemed prior to the two dietary recalls at mid- and post-intervention.
Subgroup Analyses by Child Age | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by the age of the child
Subgroup Analyses by Redemption Period | Assessed pre- and post-intervention (i.e., after participants have redeemed at least 15 weeks of coupons)
  Subgroup analyses to examine whether the impact of the intervention on primary and secondary outcomes differed by redemption period

CONTACTS AND LOCATIONS:
Overall Officials: Dana Lee Olstad, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- Participants recruited in 93 communities across British Columbia, Canada, Communities Across BC, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be available from the authors upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2026 - August 2031
Access Criteria: Data will be available from the authors upon reasonable request.

REFERENCES:
- See also: BC Farmers' Market Nutrition Coupon Program — https://bcfarmersmarket.org/coupon-program/how-it-works/